CLINICAL TRIAL: NCT04534452
Title: A Multicenter, Consumer Product Evaluation of a Single Dose of Phenylephrine Hydrochloride 30 mg Extended Release Tablets (Sinus Comfort™)
Brief Title: Study to Find Out Whether Participants With a History of Stuffy Nose Due to Allergic Reactions in the Nose Would Intend to Buy Drug Phenylephrine Hydrochloride Extended Release Tablets After Receiving it Once in This Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18146
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Nasal Congestion Due to Allergic Rhinitis
Keywords: Allergic Rhinitis with Nasal congestion
MeSH Terms: interventions — Oxymetazoline

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phenylephrine HCl (Experimental): Subjects have a documented and/or self-reported history of allergic rhinitis with nasal congestion for at least 2 years.
  Interventions: Drug: Phenylephrine HCl (Sinus Comfort, BAY112476)

INTERVENTIONS:
Drug: Phenylephrine HCl (Sinus Comfort, BAY112476) — 30 mg Extended Release Tablets, single oral dose

SUMMARY:
The researchers in this study want to find out whether participants with a history of stuffy nose due to allergic reactions in the nose would intend to buy drug Phenylephrine Hydrochloride (Phenylephrine HCl) extended release tablet (a pill is formulated so that the drug is released slowly over time) after receiving it once in this study. Phenylephrine HCl is an over-the-counter (OTC) drug (a medicine that can be bought without a prescription) used to provide temporary relief of stuffy nose caused by cold or allergies in mouth, nose and throat. Phenylephrine HCl immediate-release tablet (a pill with drug released rapidly without special rate controlling) was already approved to be used for adults and children and the recommended dose for adults and children 12 years or older is 10mg every 4 hours. Phenylephrine HCl 30mg extended release tablet used in this study is not yet approved but under development with a goal to relieve stuffy nose for every 8 hours. Researchers also want to find out if participants have any medical problems during the trial.

Participants in this study will be asked to record their stuffy nose symptoms in a diary before and after drug intake. At 8 hours after drug intake, participants need to assess whether they intends to buy the drug or not and their overall satisfaction of the stuffy nose relief. At the end the participants will complete a questionnaire about their job, learning background, income and medical history of stuffy nose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers must be 18 to 60 years old.
* Subjects must currently use or have previously used oral decongestant products.
* Subjects must have a documented and/or self-reported history (of at least 2 years) of allergic rhinitis with nasal congestion.
* Subjects must be willing to stop use of current decongestant and allergy medications during the study, and for the number of wash-out days required for their medication prior to the run-in period.
* Subjects must have nasal congestion due to allergic rhinitis of at least mild severity (sign/symptom clearly present, but minimal awareness; easily tolerated) at Visits 1 and 2.
* Subjects must have a mean seated (after 5 minutes of rest) systolic/diastolic blood pressure ≤ 138/88 mmHg.
* Subjects must have normal or clinically acceptable physical exam.
* Subjects must agree not to take monoamine oxidase inhibitor (MAOI) for 14 days before study participation and 14 days after the end of the study.
* Subjects must be willing to give written informed consent (prior to any study related procedures being performed) and able to adhere to restrictions and examination schedules.
* Female subjects of childbearing potential (a non-menopausal female who has not had a hysterectomy, bilateral oophorectomy, or medically documented ovarian failure, including a young woman who has not yet started menstruating) must be using medically acceptable (documented failure rate of less than 1%) birth control measures. Examples of medically acceptable contraception include hormonal contraceptives, intrauterine device (IUD), double-barrier method (any combination of male or female condom, diaphragm, spermicidal gel, sponge) or sterilization.

Exclusion Criteria:

* Subjects must not have any significant medical condition which, in the judgment of the investigator, is a contraindication to the use of phenylephrine HCl, might interfere with the study or requires treatment expected to affect the blood pressure. These may include thyroid disease (e.g. hyperthyroidism, hypothyroidism), uncontrolled diabetes mellitus, coronary heart disease, ischemic heart disease, elevated intraocular pressure, prostatic hypertrophy, etc.
* Subjects that have received allergen immunotherapy (if less than 3 months of stable dosing prior to screening) or Xolair (omalizumab) therapy within the past two years.
* Subjects who have a history of any clinically significant local or systemic infectious disease within four weeks prior to treatment administration.
* Subjects who have participated in a clinical trial of an investigational treatment within 30 days prior to the start of the study.
* Subjects who are, appear to be, or are known to be, current or former addicts or alcoholics.
* Subjects who have a known allergy or intolerance to phenylephrine HCl or any other decongestant, or any antihistamine.
* Females who are pregnant, nursing or unwilling to use/practice medically acceptable contraception (documented failure rate of less than 1%).
* Subjects who have used a nasal decongestant or phenylephrine-containing product other than study medication after the start of the study and during the washout period.
* Subjects with a history of asthma, rhinitis medicamentosa, or presenting with acute or chronic sinusitis.
* Subjects that have used inhaled, oral, rectal, topical (intranasal corticosteroids for allergic rhinitis are permitted), intramuscular, and/or intravenous chronic or intermittent corticosteroids (up to 1% topical hydrocortisone is permitted).
* Subject who have family or who currently or previously have been employed in the pharmaceutical industry.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 347 (Actual)
Dates: Start 2012-05-12 (Actual); Primary Completion 2012-06-06 (Actual); Study Completion 2012-06-06 (Actual)

PRIMARY OUTCOMES:
Purchase intent evaluated by using the 5-point scale | At approximately 8 hours postdose
  * 4 = Very Acceptable
  * 3 = Acceptable
  * 2 = Somewhat acceptable
  * 1 = Somewhat unacceptable
  * 0 = Very unacceptable

SECONDARY OUTCOMES:
Overall satisfaction for nasal congestion relief evaluated by using the 5-point scale | At approximately 8 hours postdose
  * 4 = Very Acceptable
  * 3 = Acceptable
  * 2 = Somewhat acceptable
  * 1 = Somewhat unacceptable
  * 0 = Very unacceptable

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Allergy & Asthma Specialists, PC, Blue Bell, Pennsylvania, United States